CLINICAL TRIAL: NCT02943005
Title: Post-operative Mobilisation After Rotator Cuff Repair: Sling Versus Nothing. A Randomized Prospective Study.
Brief Title: Post-operative Mobilisation After Rotator Cuff Repair
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: La Tour Hospital (Other)
Responsible Party: Principal Investigator, Adrien Schwitzguebel, Investigator, La Tour Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-00818
Record Dates: First submitted 2016-10-09; First posted 2016-10-24 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2016-12

CONDITIONS: Rotator Cuff

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rotator cuff repair with sling (Active Comparator): Patients wear a sling during 4 weeks, they also move passively during this period. Then progressive active mobilization is done.
  Interventions: Procedure: Rotator cuff repair
- Rotator cuff repair without sling (Experimental): Patients don't wear any sling, they move passively in all axes during 4 weeks. Then progressive active mobilization is done.
  Interventions: Procedure: Rotator cuff repair

INTERVENTIONS:
Procedure: Rotator cuff repair

SUMMARY:
The aim of this study is to compare rehabilitation with the wearing of a sling, to rehabilitation without any immobilization after an arthroscopic repair of the supraspinatus tendon. The goal is to offer to patients a simplified rehabilitation management, with a faster recovery, less pain and a quicker return to normal life.

DETAILED DESCRIPTION:
Rotator cuff tear is a frequent problem, increasing with age1. Thus arthroscopic repair is a frequent surgery. Despite this important number of cuff repair, the re-tear rate varies from 20 to 90% depending on tear severity and type of repair1,2. Many factors are implicated in tendon healing and post-operative clinical results. Some are unchangeable (age, tear size, chronicity…) but some are under the surgeon control like the surgical technique and the post-operative rehabilitation protocol. It exists many surgical repair techniques6, 7, with a massive development of technology during the last twenty years. However in terms of rehabilitation, there is only few studies and evidence of best practices4. The main aspect on which the surgeon can act, is the immobilization time. Actually, standard protocols include an immobilisation of 4 to 6 weeks before physiotherapy beginning5.

A recent review of the literature3 has highlighted five studies comparing different rehabilitation protocols, which include different immobilization periods ranging from 0 to 8 weeks, and different types of mobilization (under physiotherapist supervision or not, with machine or not). They found a similar rate of re-tear between the different protocols. But early passive motion enables to improve the range of motion during first 3-6 months, with similar results at one year.

However in all these studies, all patients had to wear a sling for at least 4 weeks, even in the early mobilization group. But the investigators don't know if this sling is really useful, probably not if the investigators follow the logic of faster recovery and same long term results with early mobilization. At our best knowledge, no study has sought to compare the usefulness of sling wearing after a rotator cuff repair. Removing sling could simplify rehabilitation and should provide a return to normal function faster, with greater satisfaction and a similar rate of re-tear.

The aim of this study is to compare rehabilitation with the wearing of a sling, to rehabilitation without any immobilization after an arthroscopic repair of the supraspinatus tendon.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old
* Small tear (< 3cm) of the supraspinatus tendon
* Arthroscopic cuff repair

Exclusion Criteria:

* Lesion of the anterior or posterior rotator cuff
* Significant other trauma of the involved upper member (e.g. associated scapular or clavicular fractures, acromioclavicular dislocation)
* Preoperative shoulder stiffness
* Inability to follow properly post-surgery recommendations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
ASES score | 3 months
  Clinical score (0-100)

SECONDARY OUTCOMES:
Retear or non healing of the rotator cuff | 6 months
  Ultrasound control

OTHER OUTCOMES:
Return to sports | 6 months
  Yes/no
Work absenteeism | 6 months
  Months
Complications (i.e frozen shoulder) | 6 months
  Description of complication
Number of physiotherapy sessions needed. | 6 months
  Clinical evolution
VAS score | 1.5, 3, and 6 months
  Graded between 0 and 10
Constant score | 1.5, 3, and 6 months
  Clinical scores number between 0-100
SANE score | 1.5, 3, and 6 months
  Clinical scores number between 0-10
ASES score | 1.5, 3, and 6 months
  Clinical scores number between 0-100
Strength of arms in Jobe position | 6 months
  Strength measurement in kilo according to the technique of Int Shoulder Surg Collin et al. In press

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Lädermann, MD, Principal Investigator — La Tour Hospital
Locations (1):
- La Tour Hospital, Meyrin, Canton of Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No